CLINICAL TRIAL: NCT00709085
Title: Functional Genomics and Proteomics Towards and Understanding of Cell Signaling and Diseases--- Genomic and Proteomic Analyses of Liver Cells During Hepatitis Virus Infections and Cell Therapy (4/4)
Brief Title: To Study the Effects of Host Genetic Factors on Liver Cirrhosis and Hepatocellular Carcinoma (HCC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Ming-Fu Chang, Ph.D., Proferrsor, Institute of Biochemistry and Molecular Biology, National Taiwan University
Other Study IDs: 200803038R
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Liver Cirrhosis
Keywords: single nucleotide polymorphism
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — liver tissue (non-tumor part)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: HCC patients without liver cirrhosis
- 2: HCC patients with liver cirrhosis

SUMMARY:
The purpose of this study is to identify genetic determinants of susceptibility to liver cirrhosis and hepatocellular carcinoma. It will assist in predicting individual risks of disease progression and would help to clarify pathophysiologic mechanisms of liver cirrhosis and hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) usually occurs in cirrhotic liver. Only 10-30% of HCC occur in non-cirrhotic liver. It has been suggested that etiological factors may differ for HCC which develop in cirrhotic liver: HCC in non-cirrhotic liver might be less often associated with viral infection and chronic alcoholism than HCC in cirrhotic livers. However, in any individual, the factors that determine HCC with or without cirrhosis remain unknown.

Cirrhosis is the end of fibrosis progression. The progress of liver fibrosis is a complex progress involving many cytokines related to activation of the hepatic stellate cells and progressive accumulation of extracellular matrix. The key enzymes responsible for deposition and degradation of all the protein component of extracellular matrix and basement membrane are matrix metalloproteinases.

To assess whether genetic variations in cytokines and matrix metalloproteinases result in diversity of liver cirrhosis and HCC, we conduct a case-control study of single nucleotide polymorphism analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatocellular carcinoma
* restrict the casual agent of liver disease to viral infection

Exclusion criteria:

* the casual aget of liver disease is not viral infection, such as alcohol abuse

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 596 patients with histologically proven HCC were collected by Dr. Po-Huang Lee's Lab. (The Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan)
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Fu Chang, Ph.D., Study Chair — National Taiwan University College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan